CLINICAL TRIAL: NCT02419066
Title: Examining HIV Treatment Adherence During Early Disease
Acronym: META
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Mbarara University of Science and Technology (Other); Desmond Tutu HIV Centre (Other)
Responsible Party: Principal Investigator, Jessica Haberer, MD, Dr. Jessica Haberer, MD, MS, Massachusetts General Hospital
Other Study IDs: OPP1113634
Record Dates: First submitted 2015-04-06; First posted 2015-04-17 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Medication Adherence; HIV
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — plasma, dried blood spots
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- men and women with CD4 >=350: electronic monitoring of ARV adherence in men and women with CD4 >=350
- pregnant women with CD4 >=350: electronic monitoring of ARV adherence in pregnant women with CD4 >=350
- men and women with CD4 <200: electronic monitoring of ARV adherence in men and women with CD4 <200

SUMMARY:
Determine the level, patterns, and correlates of objectively measured ART adherence in early and advanced-stage disease, among pregnant and non-pregnant individuals, to determine the need and nature of interventions to support early ART adherence in Uganda and South Africa

DETAILED DESCRIPTION:
Specific Aims

Aim 1: Determine the level, patterns, and correlates of objectively measured ART adherence in early and advanced-stage disease, among pregnant and non-pregnant individuals, to determine the need and nature of interventions to support early ART adherence in Uganda and South Africa. Outcomes include: i) average adherence, ii) incidence of any 28-day period with <80% adherence, iii) number of ART interruptions >72 hours (which could lead to loss of viral suppression), and iv) detectable HIV RNA >400 copies/Ml at 6 and 12 months. Guided by prior work and the Theory of Vulnerable Populations, we hypothesize that incomplete adherence will be associated with a) early-stage, asymptomatic disease, b) pregnancy and postpartum periods, and c) multiple social and economic factors. Individuals with CD4 200-350 will not be studied in order to most efficiently identify differences at the extremes of early and advanced disease.

Aim 2: Given the known importance of social networks and social support for adherence in advanced-stage disease in some RLS, we will determine the extent to which social network cohesion, HIV serostatus disclosure within the network, and receipt of social support explain differential ART adherence in early and advanced-stage disease. We hypothesize that: i) compared to people with advanced-stage disease, people with early-stage disease will have less cohesive social networks, disclose their seropositivity to fewer network members, and receive less social support; ii) social network cohesion, serostatus disclosure, and social support will be associated with greater ART adherence; and iii) these associations will explain a significant portion of differential ART adherence in early versus advanced-stage disease. Additionally, although these factors have been well established previously in Uganda, prospective data is needed to account for secular trends related to treatment expansion and comparable data are needed from South Africa.

Aim 3: We will use qualitative methods to identify, describe and explain influences on ART adherence in early-stage disease to guide intervention development. In-depth understanding of influences on ART adherence among individuals with early-stage HIV disease will inform the focus of any needed ART adherence interventions for this population. We will conduct in-depth, adherence-focused qualitative interviews with (a) 50 HIV+ men and non-pregnant women, and (b) 50 HIV+ pregnant women, who initiate ART with early-stage disease. Interviews with pregnant women may be post-partum by the time of the interview. Equal numbers of individuals in these two groups will be drawn from the Uganda and South Africa sites.

Study Procedures

Aims 1, 2:

Upon recruitment, participants will receive a baseline interview and phlebotomy. Women <50 years will be given a urine pregnancy test. Participants will be given a Wisepill device, and instructed on how to use it using training procedures established in prior studies by this group. The RA will then fill the Wisepill device with the antiretroviral medication. If feasible and acceptable to participants, participants will then be driven to their place of residence for global positioning system (GPS) mapping (given that GPS-measured distance has been associated with clinic visit adherence). If available, existing GPS map data may be used in lieu of driving to the participant's place of residence and collecting GPS coordinates. Structured interviews will be conducted at enrollment, 6 and 12 months. Interviews will typically take place at the clinic. If feasible and desirable, they may be offered at home or another location of the participant's choosing. It will be explained clearly to the participant that if they do not have adequate cellular reception for reliable data transmission via the Wisepill device they need to bring the Wisepill device to clinic for pharmacy refill will be emphasized. Additionally, if they permanently move to an area that is more than 60 km from the clinic, they will be disenrolled from the study.

The 6 and 12-month follow up visits will be held separately from routine clinic visits to avoid potential influence on routine clinic attendance and/or adherence (e.g., easier transportation or higher motivation to attend due to study visit incentives). Participants may be sought by phone or at home for study procedures if they do not attend their scheduled 6 and 12-month clinic visits. Individuals may also be contacted if the study team becomes aware of technical problems with the Wisepill device. In that event, the study team will try to reach the participant by phone, but if they are unable, they may go to the participant's house to assess the technical difficulties.

As noted above, participants will be seen at baseline, 6 months, and 12 months for structured interviews, phlebotomy (viral load, sample storage), and for women, pregnancy testing. Because of the dynamic relationship between adherence and HIV RNA suppression, the first year is the most critical period for adherence and because the greatest decline in adherence is usually seen over the first year, a full year of observation is planned to determine if stage of disease is associated with adherence.

Structured interviews will cover the following topics: demographics, health status, socio-economic status, structural barriers to clinic access, food security, physical and mental health, depression, coping, sexual behavior, transactional sex/intimate partner violence, beliefs/satisfaction, necessity/concerns, alcohol and recreational drug use, stigma, adherence, and medical mistrust/conspiracy. We will also define social networks.

Adherence will be measured in real-time with the Wisepill device, which automatically captures and reports, once daily via cellular technology, the participant's medication adherence data. A second signal is transmitted daily to report battery level and confirm device functionality.

Aim 3:

We will use purposeful sampling to systematically represent subgroups of early disease adherers (both low and high) and create the conditions for in-depth qualitative analysis. Starting at 6 months of follow-up, we will identify from the larger cohorts of participants, 25 pregnant early disease adherers and 25 non-pregnant early disease adherers at each of the two (Ugandan and South African) study sites (total qualitative sample size = 100 individuals). Interviews with pregnant women may occur during the post-partum period. Each qualitative participant will take part in a single, in-depth individual interview conducted by a research assistant trained in the collection of in depth qualitative interviews. Interviews will target the actual adherence experiences and behavior of interviewees and systematically cover a range of relevant topics, including: (a) the circumstances under which pills are taken (dosing behavior); (2) missed doses and why they happened; (3) what obstacles impede adherence; (3) who helps with adherence and how (social support). Interviews will be transcribed into English, if needed, to produce the qualitative data set of 100 interview transcripts.

ELIGIBILITY:
Inclusion Criteria:

* • Participants will be ART naïve and initiating within one month of enrollment date

  * Participants will be at least 18 years of age
  * Participants will be able to provide informed consent
  * Participants will live within 60 km of the clinic; intention to stay in the area for the next year
  * Participants will either be 1) in early-stage disease (CD4>350) with WHO stage I (i.e., asymptomatic), or 2) in advanced-stage disease (CD4<200).
  * Pregnant participants will be 34 weeks or less in pregnancy (per best available estimates

Exclusion Criteria:

* • Live >60 km from the clinic (due to logistics of following participants) or intention to move outside 60km area within the next year

  * <18 years old (adherence patterns and determinants likely differ significantly from those >18 years)
  * Currently in an intermediate stages of disease (i.e., CD4 200-349; the intent of the proposed research is to examine differences in adherence between HIV-infected people initiating ART at early versus advanced-staged disease)
  * Women who have a CD4<200 and who report current pregnancy at the time of consent
  * Unable to provide informed consent (e.g., due to mental limitations or intoxication)
  * Anyone who does not initiate on ART within 1 month of the enrollment date
  * Any pregnant participant greater than 34 weeks in pregnancy (per best available estimate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be HIV-infected adults initiating antiretroviral therapy at recruitment sites in southwestern Uganda (Mbarara, Kabwohe) and Cape Town (Gugulethu) South Africa. They will have either early (CD4 >350) or late (CD4 <200) HIV infection.
Sampling Method: Non-Probability Sample
Enrollment: 904 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
HIV Adherence | 12 months
  ART adherence will be monitored continuously, up to 12 months, using the Wisepill device.

SECONDARY OUTCOMES:
HIV RNA viral load | 12 months
  Colleced at 12 months after ART initiation and categorized as a binary variable at the later time points: Undetectable (<400 copies/mL) vs. detectable (greater than equal to 400 copies/mL)
Retention in HIV care | Attendance at scheduled visit (w/in 45 days)
  Defined as attendance (within 45 days) at scheduled appointments after initiation of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Haberer, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- Hannan Crusaid Treatment Centre (HCTC), Gugulethu, Cape Town, Western Cape, South Africa
- Immune Suppression Syndrome (ISS) Clinic, Mbarara, Mbarara District, Uganda

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available at the end of the study upon request.